CLINICAL TRIAL: NCT06850597
Title: Randomized, Double-blind, Placebo- Controlled Trial Evaluating Efficacy and Safety of Dimethyl Fumarate in Brain Atrophy Reduction, Synaptic Functional Connectivity, Cognitive Functions, Quality of Life, and Activity of Daily Living Improvement Among Patients with Mild Cognitive Impairment and Dementia Due to Alzheimer's Disease
Brief Title: Efficacy and Safety of Dimethyl Fumarate Among Patients with Mild Cognitive Impairment and Dementia Due to Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jakub Kazmierski, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010622; 2022-002171-11 (EudraCT Number)
Record Dates: First submitted 2024-12-09; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: MCI; MCI-AD, Early Stage Alzheimer's Disease; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Assessment of the degree of improvement in cognitive functions in diagnosed patients MCI and AD. (Placebo Comparator): Assessment of the degree of improvement in cognitive functions, including memory, attention, thinking, executive and language functions in diagnosed patients MCI and AD taking dimethyl fumarate 480 mg daily compared to patients taking placebo.
  Interventions: Drug: dimethyl fumarate
- Assessment of the safety of therapy (Other): Assessment of the safety of therapy
  Interventions: Drug: dimethyl fumarate
- Assessment of the impact of therapy on patients' daily functioning (Placebo Comparator): Assessment of the impact of therapy on patients' daily functioning - Scale Alzheimer's Disease Cooperative Study - Activity of Daily Living (ADCS-ADL).
  Interventions: Drug: dimethyl fumarate
- Assessment of the impact of therapy on the presence of symptoms neuropsychiatric/behavioral disorder (Placebo Comparator): Assessment of the impact of therapy on the presence of symptoms neuropsychiatric/behavioral disorders in patients scale Neuropsychiatric Inventory (NPI), Geriatric Depression Scale (GDS).
  Interventions: Drug: dimethyl fumarate
- Assessment of the impact of therapy on the quality of life of patients and their caregivers (Placebo Comparator): Assessment of the impact of therapy on the quality of life of patients and their caregivers (scales EQ-5D; Zarit Burden Interview).
- reducing the degree of brain atrophy in patients - MRI examination (Placebo Comparator): Assessment of the impact of therapy on reducing the degree of brain atrophy in patients from the active group compared to the control group (MRI examination)
  Interventions: Drug: dimethyl fumarate
- impact of therapy on improvement in functional connections assessed in rs-fMRI rs-EEG (Placebo Comparator): Assessment of the impact of therapy on improvement in functional connections assessed in rs-fMRI and rs-EEG
  Interventions: Drug: dimethyl fumarate
- Effect of therapy on peripheral markers of oxidative stress and pro-inflammatory markers (Placebo Comparator): Assessment of the effect of therapy on peripheral markers of oxidative stress and pro-inflammatory markers
  Interventions: Drug: dimethyl fumarate
- degree of reduction in the rate of progression from MCI to dementia after completion (Placebo Comparator): Assesment of the degree of reduction in the rate of progression from MCI to dementia after completion of the clinical phase of the study
  Interventions: Drug: dimethyl fumarate
- degree of improvement in cognitive functions using the MMSE and CDR scales (Placebo Comparator): Assessment of the degree of improvement in cognitive functions using the MMSE and CDR scales
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — 480 mg per day
  Arms: Assessment of the degree of improvement in cognitive functions in diagnosed patients MCI and AD.; Assessment of the impact of therapy on patients' daily functioning; Assessment of the impact of therapy on the presence of symptoms neuropsychiatric/behavioral disorder; Assessment of the safety of therapy; Effect of therapy on peripheral markers of oxidative stress and pro-inflammatory markers; degree of improvement in cognitive functions using the MMSE and CDR scales; degree of reduction in the rate of progression from MCI to dementia after completion; impact of therapy on improvement in functional connections assessed in rs-fMRI rs-EEG; reducing the degree of brain atrophy in patients - MRI examination

SUMMARY:
The goal of this clinical trial is to assess the degree of improvement in cognitive functions, including memory, attention, thinking, executive and language functions in diagnosed patients MCI and AD taking dimethyl fumarate 480 mg daily compared to patients taking placebo. Participant will be 55 to 90 years old, both genders. The main question it aims to answer is: Changing the degree of cognitive improvement based on the RBANS score among patients diagnosed with MCI and AD after completing dimethyl fumarate therapy test group compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 55-90 years.
2. Patients diagnosed with mild cognitive impairment in Alzheimer's disease and mild to moderate Alzheimer's dementia (MMSE >16) diagnosed based on NIA-AA criteria.
3. MMSE score from 17 to 30 points.
4. CDR score from 0.5 to 2.
5. The patient signs an informed, voluntary consent to participate in the study.
6. The patient has a close person/de facto guardian who agrees to help the patient during participation in the study.
7. At least 6 years of education.
8. In the case of anti-Alzheimer's drugs, the use of cholinesterase inhibitors is permitted provided that they are included at least 3 months before entering the study and used at a stable dose for at least 60 days before entering the study. In the case of memantine, its use is permitted provided that it is included at least 4 months before entering the study and used at a stable dose for at least 3 months before entering the study.

Exclusion Criteria:

1. Lack of informed voluntary consent to participate in the study.
2. Patients who cannot read or write.
3. Pregnant, breastfeeding or childbearing women who do not use effective contraception (hormonal contraception, surgical sterilization, intrauterine device, condom in combination with vaginal spermicide).
4. Participation in another clinical trial, currently or within 3 months prior to the screening visit.
5. Liver failure (i.e. cirrhosis or active liver disease), diagnosed acute or chronic hepatitis regardless of cause.
6. Chronic kidney disease with GFR below < 60 ml/min/m2
7. Abnormal liver parameters: ALAT exceeding > 2 times the upper limit of normal
8. Leukopenia (<4000/mm3), granulocytopenia (<1500/mm3) or lymphopenia (<1000/mm3) regardless of the cause.
9. Severe agitation.
10. Mental retardation.
11. Delirium diagnosed according to DSM-5 criteria.
12. Diagnosis of neurological and neurodegenerative diseases other than Alzheimer's disease (multiple sclerosis, Parkinson's disease, Huntington's disease, previous stroke).
13. Presence of hemorrhagic foci in magnetic resonance imaging with a diameter of ≥ 2 cm3, more than three (3) ischemic stroke foci with a diameter of ≥ 1.5 cm3 or a single ischemic foci with a diameter of ≥ 2 cm3, presence of vascular malformations, aneurysms, subdural hematoma, normal pressure hydrocephalus, final decision at the discretion of the investigator.
14. Severe or uncontrolled somatic disease that could affect the course of the study (e.g. neoplastic, cardiovascular, respiratory, metabolic or digestive, severe renal failure, unstable type I or II diabetes, untreated or uncontrolled clinically significant hypertension).
15. Use of benzodiazepines or barbiturates within 1 week prior to screening.
16. Pharmacological immunosuppression.
17. Patients with bipolar disorder or psychotic disorders or any other psychiatric condition (current or past) that the Investigator believes interferes with the study.
18. Alcoholism or drug addiction as defined by DSM-5 within the past 5 years (dependent for more than 1 year and or in remission for less than 3 years).
19. Patients with any medical condition that, in the Investigator's judgment, is an exclusion criterion.
20. Thyroid hormone therapy initiated, discontinued, or modified within 3 months prior to screening visit.
21. Menopausal hormone replacement therapy initiated, discontinued, or modified within 3 months prior to screening visit.
22. Use of prohibited drugs in the study: Antineoplastic drugs (no studies). Immunosuppressive drugs (no studies). Corticosteroids (impact on project results). Live attenuated vaccines (no studies). Inactivated vaccines may be used. Benzodiazepines (impact on assessed endpoints). Other ethyl esters used orally or topically.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the degree of cognitive improvement based on the RBANS score among patients diagnosed with MCI and AD after completing dimethyl fumarate therapy test group compared to the placebo group. | 15 months
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a neuropsychological measure used in the assessment of cognitive function in older adults, studies of mild cognitive impairment and Alzheimer's disease dementia, and studies evaluating the effectiveness of therapeutic interventions. The test generates index scores in five neurocognitive domains, as well as a Total Scale Index score. The RBANS is characterized by high sensitivity in detecting disease and assessing changes in scores during treatment in patients with MCI in the course of Alzheimer's disease. with MCI and AD after completing dimethyl fumarate therapy test group compared to the placebo group.

SECONDARY OUTCOMES:
Assessment of the safety of therapy | 15 months
Assessment of the impact of therapy on the daily functioning of patients - Alzheimer's Disease Cooperative Study - Activity of Daily Living (ADCS-ADL) scale. | 15 months
Assessment of the impact of therapy on the presence of neuropsychiatric symptoms/behavioral disorders in patients using the Neuropsychiatric Inventory (NPI) scale and the Geriatric Depression Scale (GDS). | 15 months
Assessment of the impact of therapy on the quality of life of patients and their caregivers (EQ-5D scales; Zarit Burden Interview). | 12 months
Assessment of the effect of therapy on the reduction of the degree of brain atrophy in patients from the active group compared to the control group (MRI study). | 6 months
Assessment of the effect of therapy on the improvement of functional connections assessed in rs-fMRI and rs-EEG. | 15 months
  EEG and MRI data will be processed using standard processing pipelines. The results will be a topographic map of the EEG frequency band distribution on the brain surface, temporal and time-frequency analyses based on FFT and wavelets, entropy analysis, and EEG coherence markers. Then, inverse localization of EEG signals generated on the scalp over the brain surface will be performed. Particular emphasis will be put on frontal structures and areas detected by MRI clustering. We will perform machine learning-based clustering of EEG and MRI data to detect significant features.
  CDR "Clinical Dementia Rating Assessment" score from 0.5 to 2

OTHER OUTCOMES:
Assessment of the effect of therapy on peripheral markers of oxidative stress and pro-inflammatory markers. | 6 months
Assessment of the degree of reduction of the MCI progression rate to dementia after the end of the clinical phase of the study. | 12 months
Assessment of the degree of improvement of cognitive functions using the MMSE and CDR scales. | 15 months
  MMSE (Mini-Mental State Examination) score from 17 to 30 points CDR (The Clinical Dementia Rating) score from 0,5 to 2 points

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Old Age Psychiatry and Psychotic Disorders Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No